CLINICAL TRIAL: NCT04630483
Title: The Effect of Different Anesthesia Methods on the Platelet-lymphocyte and Neutrophil-lymphocyte Ratio in Patients Undergoing Cancer Surgery
Brief Title: Platelet-lymphocyte and Neutrophil-lymphocyte Ratio in Patients Undergoing Cancer Surgery
Status: Withdrawn | Type: Observational
Why Stopped: No participants
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Bahadir Ciftci, Principal Investigator, Medipol University
Other Study IDs: Medipol Hospital 17
Record Dates: First submitted 2020-11-10; First posted 2020-11-16 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Cancer; Urologic Neoplasms; Gynecologic Cancer
Keywords: Cancer surgery; Anesthesia; Neutrophil-to-lymphocyte ratio; Platelet-to-lymphocyte ratio
MeSH Terms: conditions — Neoplasms; Urologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I: INHA: Inhalational anesthesia (INHA)
  Interventions: Other: INHA
- Group II: TIVA: Total intravenous anesthesia (TIVA)
  Interventions: Other: TIVA

INTERVENTIONS:
Other: INHA — NLR and PLR ratio will be assessed at postoperative 6th and 24th hours compared to preoperative values
  Groups: Group I: INHA
Other: TIVA — NLR and PLR ratio will be assessed at postoperative 6th and 24th hours compared to preoperative values
  Groups: Group II: TIVA

SUMMARY:
Cancer is a major cause of morbidity and mortality worldwide. Despite the use of surgery in an attempt to cure the majority of solid tumors, metastasis from residual cancer cells still remains a major cause of morbidity and mortality. General anesthesia and surgical stress during surgery suppress the immune response by directly affecting the immune system or by activating the hypothalamic-pituitaryadrenal axis and the sympathetic nervous system. The aim of our prospective observational study was to assess the value of neutrophil-to-lymphocyte ratio and platelet-to-lymphocyte ratio regarding outcome underwent cancer surgery. Primary aim is to assess the preoperative and postoperative values of inhalational anesthesia vs total intravenous anesthesia.

DETAILED DESCRIPTION:
Cancer is a major cause of morbidity and mortality worldwide. Despite the use of surgery in an attempt to cure the majority of solid tumors, metastasis from residual cancer cells still remains a major cause of morbidity and mortality. As is the case with most cancers, loco-regional recurrence and distant metastases are all too common, even after successful surgical treatment and adjuvant therapy. Cancer metastasis is a complex process in which cancer cells evade the immune system. Cancer cells gain the ability to proliferate, migrate, and invade adjacent tissues, and together with angiogenesis, these capabilities facilitate the successful metastasis of cancer.

General anesthesia and surgical stress during surgery suppress the immune response by directly affecting the immune system or by activating the hypothalamic-pituitaryadrenal axis and the sympathetic nervous system. Along with surgical stress, blood transfusion, hypothermia, and postoperative pain, anesthetics are associated with immunosuppression during perioperative periods because anesthetics/analgesics have direct suppressive effects on cellular and humoral immunity. In general anesthesia, it is suggested that inhalational anesthesia (INHA) such as sevoflurane and isoflurane may modulate antimetastatic immunity by inhibiting NK cell cytotoxicity and inhibit T helper cell proliferation. This could potentially be unfavorable for cancer survival. In contrast, propofol-based total intravenous anesthesia (TIVA) is suggested to have anti-inflammatory features and to be advantageous compared with INHA by promoting the activation of T-helper cells, decreasing matrix metalloproteinases, and not suppressing NK cell activity to the same extend as INHA. The immunological impact of the anesthetic agents may thus influence clinical measures including overall mortality and postoperative recovery. Recently, some readily available parameters, originated from routine complete blood count (CBC), have been investigated as potential biomarkers with mixed results and no consensus so far regarding its accuracy and clinical usefulness: neutrophil-to-lymphocyte ratio (NLR), monocyte-to lymphocyte ratio (MLR), platelet-to-lymphocyte ratio (PLR), and mean platelet volume-to-platelet count (MPV/PC) ratio.

The aim of our prospective observational study was to assess the value of NLR and PLR ratio regarding outcome underwent cancer surgery. Primary aim is to assess the preoperative and postoperative values of inhalational anesthesia vs total intravenous anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I-II
* Scheduled for elective cancer surgery (urology, general surgery, gynecologic) under general anesthesia

Exclusion Criteria:

* Secondary sepsis and/or septic shock with an underlying condition
* Active infection such as severe peritonitis, pancreatitis, or trauma
* Long-term ICU stay
* Preexisting immunodeficiency.

Ages: 20 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Scheduled for elective cancer surgery (urology, general surgery, gynecologic)
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
The value of NLR and PLR ratio | Average 6 months, through study completion
  Primary aim is to assess the preoperative and postoperative values of inhalational anesthesia vs total intravenous anesthesia.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We will not plan to share IPD

REFERENCES:
- [Background] Kim R. Anesthetic technique and cancer recurrence in oncologic surgery: unraveling the puzzle. Cancer Metastasis Rev. 2017 Mar;36(1):159-177. doi: 10.1007/s10555-016-9647-8. PMID 27866303
- [Background] Kim R. Effects of surgery and anesthetic choice on immunosuppression and cancer recurrence. J Transl Med. 2018 Jan 18;16(1):8. doi: 10.1186/s12967-018-1389-7. PMID 29347949
- [Background] Djordjevic D, Rondovic G, Surbatovic M, Stanojevic I, Udovicic I, Andjelic T, Zeba S, Milosavljevic S, Stankovic N, Abazovic D, Jevdjic J, Vojvodic D. Neutrophil-to-Lymphocyte Ratio, Monocyte-to-Lymphocyte Ratio, Platelet-to-Lymphocyte Ratio, and Mean Platelet Volume-to-Platelet Count Ratio as Biomarkers in Critically Ill and Injured Patients: Which Ratio to Choose to Predict Outcome and Nature of Bacteremia? Mediators Inflamm. 2018 Jul 15;2018:3758068. doi: 10.1155/2018/3758068. eCollection 2018. PMID 30116146